CLINICAL TRIAL: NCT04269993
Title: Impact of Acute Cannabis Administration on Pain Symptomology and Inflammatory Markers Among Patients With Rheumatoid or Psoriatic Arthritis
Brief Title: Impact of Cannabis on Pain and Inflammation Among Patients With Rheumatoid or Psoriatic Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Termination of study funding
Sponsor: Brown University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Elizabeth Aston, Assistant Professor, Brown University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: #1904002430; P20GM130414 (NIH)
Record Dates: First submitted 2020-02-12; First posted 2020-02-17 (Actual); Results first posted 2025-03-13 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Rheumatoid Arthritis; Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis, Psoriatic | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vaporized cannabis: Placebo then Active THC (Experimental): Participants are randomized to receive placebo cannabis during Session 1 and Active THC cannabis during Session 2; sessions will be separated by at least 2 days
  Interventions: Drug: Cannabis: placebo and medium THC/medium CBD
- Vaporized cannabis: Active THC then Placebo (Experimental): Participants are randomized to receive Active THC cannabis during Session 1 and placebo cannabis during Session 2; sessions will be separated by at least 2 days
  Interventions: Drug: Cannabis: placebo and medium THC/medium CBD

INTERVENTIONS:
Drug: Cannabis: placebo and medium THC/medium CBD — Vaporized cannabis was administered to participants (placebo and medium THC/medium CBD).
  Other Names: Marijuana

SUMMARY:
This laboratory study will investigate the impact of cannabis on pain, affect, and inflammation among patients with rheumatoid or psoriatic arthritis (n = 76). Two cannabis formulations varying in potency will be administered via vaporization across two experimental sessions using a counter-balanced, double-blind, crossover design.

DETAILED DESCRIPTION:
This laboratory study will investigate the impact of cannabis on pain, affect, and inflammation among patients with rheumatoid or psoriatic arthritis (n = 76). Two cannabis formulations varying in potency will be administered via vaporization across two experimental sessions using a counter-balanced, double-blind, crossover design. Blood will be collected during each session (pre-vaporization, 10 minutes post-vaporization, 60 minutes post-vaporization). Self-reported pain and affect will be assessed at the same time points. The effect of cannabis on pain, affect, and inflammatory biomarkers will be assessed. The study will recruit 76 patients to obtain a final sample of 66 with complete data (15% attrition). This study will be the first to investigate the effect of cannabis on pain, affect, and markers of inflammation among patients with rheumatoid or psoriatic arthritis. This study has the potential to guide clinical decisions pertaining to use of cannabis to treat arthritis symptoms with more precise recommendations regarding cannabis formulation.

ELIGIBILITY:
Inclusion Criteria:

1. current RA or PA diagnosis with active arthritis not adequately controlled by standard medication
2. if taking prescribed steroid, non-steroidal anti-inflammatory (NSAID), and/or disease-modifying anti-rheumatic drug (DMARDS; e.g., tumor necrosis factor inhibitors), must be stable use for at least 1 month prior to enrollment (all must be maintained throughout the study)
3. English-speaking or Spanish-speaking
4. negative urine toxicology screen
5. negative pregnancy test
6. not nursing
7. use of highly effective birth control during the study for both males and females
8. prior history of vaping or smoking cannabis

   Exclusion Criteria:
9. greater than zero breath alcohol concentration
10. presence of psychosis, panic disorder, or suicidal ideation or intent
11. self-report of serious adverse reaction to cannabis in the past year
12. smoking more than 20 tobacco cigarettes per day
13. body mass index below 18.0 or above 33.0 kg/m2 range confirmed during medical exam
14. all current asthma conditions (i.e., active symptomatic asthma within the last week) or current or past history of asthma triggered by smoking or vaping
15. current diagnosis of dementia or Parkinson's disease
16. below cut-off on mental status exam
17. current diagnosis of moderate to severe traumatic brain injury
18. current diagnosis of epilepsy
19. individuals who are immunocompromised (i.e., post-organ transplant, those with an immune deficiency disorder such as HIV, individuals taking immunosuppressant steroids such as continuous prednisone use, and those with lupus)
20. past kidney disease (e.g., glomerular nephritis, polycystic kidney disease) and/or presence of elevated creatinine
21. cardiac disease confirmed via clinically significant abnormal findings on an EKG (e.g., arrhythmia, conduction abnormalities, ischemia, or evidence of past myocardial infarction), as well as diagnoses of congestive heart failure or cardiomyopathy
22. abnormal vital signs
23. taking any exclusionary medications
24. presence of any severe cardiovascular, renal, or hepatic disorder
25. below 18 or above 65 years of age
26. use of cannabis in the past 1 month before commencement of study participation and throughout the study as confirmed via urine toxicology screening aa) below minimum self-reported pain level on a visual analog scale (VAS) pre-study enrollment via telephone and at baseline due to potential variability in pain level

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Aston, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University School of Public Health, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vaporized Cannabis: Placebo Then Active THC | Vaporized Cannabis: Active THC Then Placebo
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaporized Cannabis: Placebo Then Active THC | Vaporized Cannabis: Active THC Then Placebo | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 23 | 57 (1.41) | 45.67 (19.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Subjective Pain Level Post-vaporization
Description: Short-Form McGill Pain Questionnaire (SF-MPQ) Scale range to describe current pain level: 0 'none' to 10 'worst possible'
  *higher scores indicate more severe pain
Time Frame: at the termination of the cannabis administration procedure (10 minutes post-completion of cannabis administration)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vaporized Cannabis: Placebo Then Active THC | Vaporized Cannabis: Active THC Then Placebo
Number analyzed (Participants) | 1 | 2
score on a scale
  Placebo Dose | 3 | 2 (1.414)
  Medium THC/Medium CBD Dose | 4 | 4.5 (2.121)
Statistical Analysis 1: Comparison: Vaporized Cannabis: Placebo Then Active THC; Test type: Superiority; p = 0.04, t-test, 1 sided; Mean Difference (Final Values) = -2

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse events are reported per intervention (THC, Placebo)
Groups:
- Placebo: Participants receive placebo cannabis during one session; sessions will be separated by at least 2 days
- Active THC: Participants receive active THC cannabis during one session; sessions will be separated by at least 2 days
Arm/Group | Placebo | Active THC
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/93/NCT04269993/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/93/NCT04269993/ICF_001.pdf